CLINICAL TRIAL: NCT00031512
Title: A Double-Blind, Placebo-Controlled, Virologic Efficacy Trial of Pleconaril in the Treatment of Neonates With Enteroviral Sepsis Syndrome
Brief Title: Pleconaril Enteroviral Sepsis Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 99-018
Record Dates: First submitted 2002-03-06; First posted 2002-03-07 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2012-08-09

CONDITIONS: Enterovirus Infection
Keywords: enteroviral sepsis; enterovirus; infants; Pleconaril
MeSH Terms: conditions — Enterovirus Infections | interventions — pleconaril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo.
  Interventions: Other: Placebo
- Pleconaril (VP63843) (Experimental): The first dosing cohort received 5 mg/kg/dose oral every 8 hours for 7 days (21 doses) of a 40 mg/mL oral liquid formulation. Subsequent dosing cohorts are receiving 8.5 mg/kg/dose oral every 8 hours for 7 days (21 doses) of a 40 mg/mL oral suspension formulation.
  Interventions: Drug: Pleconaril

INTERVENTIONS:
Other: Placebo — Placebo.
  Arms: Placebo
Drug: Pleconaril — 5 mg/kg /dose oral every 8 hours for 7 days (21 doses) of a 40 mg/mL oral liquid formulation and 8.5 mg/kg/dose oral every 8 hours for 7 days (21 doses) of a 40 mg/mL oral suspension formulation.
  Arms: Pleconaril (VP63843)

SUMMARY:
A common group of viruses that infect humans are enteroviruses. Enteroviruses produce illnesses in children which may range from very mild (summer colds) to severe (infections of the brain, liver, and heart). The purpose of this study is to determine if a new drug called pleconaril helps treat babies with enteroviral sepsis. In addition, researchers are attempting to determine a safe and effective dose of pleconaril to help babies with this disease. Infants who are 15 days or younger when diagnosed with enteroviral disease are eligible for this study. Two out of 3 babies will be randomly assigned to receive Pleconaril and the other one out of three will receive a placebo (inactive substitute). Participants will be hospitalized while receiving study medication. Babies will receive standard treatment care for their symptoms and will be observed for their medical progress. Participants may be in the study for up to 2 years.

DETAILED DESCRIPTION:
Enteroviral infection is a serious health problem in the newborn infant. Approximately 60-70% of infants diagnosed with enteroviral disease within the first 10 days of life acquire their infection by transmission from the mother at the time of delivery. Congenital infection is rare but often fatal. Perinatal transmission of enteroviral infections in newborn nurseries has also been implicated as an important route of spread of the disease in newborn infants and postnatal transmission of enteroviral infections during seasonal peaks of enterovirus activity occurs commonly. Thus, during periods of high prevalence of enterovirus infection in the community, there are many potential sources of infection both during and after discharge from the nursery, including the mother, other family members, and hospital staff. Approximately 75% of cases of neonatal enteroviral disease carry a benign outcome, with diagnosis and symptomatic treatment in non-intensive care unit settings. For the remainder of patients, more serious consequences can result from systemic enteroviral infection, including meningoencephalitis, cardiovascular collapse, myocarditis, or hepatitis. These last two organ-specific complications carry high mortality rates. Historically, symptom management and supportive care have been the rule in the management of these patients. No specific therapeutic intervention is currently available for the management of these gravely ill neonates. The current study will evaluate the antiviral drug pleconaril as a treatment for enterovial sepsis syndrome. This trial is a multi-center, randomized, placebo-controlled study to evaluate the virologic efficacy, safety, and pharmacokinetics of pleconaril in the treatment of severe enteroviral sepsis syndrome. Patients will be randomized 2:1 to drug or placebo. For enrollment into this trial, infants must have evidence of severe hepatic involvement, myocardial involvement, and/or consumptive coagulopathy. Their age must be 15 days or less at the time of the onset of disease symptoms. Enrollment will continue until 45 subjects with confirmed enteroviral disease have been enrolled. The primary objective of this investigation is to determine if administration of pleconaril to critically ill neonates with enteroviral sepsis syndrome results in more rapid clearance of virus from various body sites. Other objectives of this study are to assess the safety and pharmacokinetics of this drug in this patient population. The effects of pleconaril on measures of clinical outcome also will be evaluated. These include the degree of inotropic and blood product support required during the acute illness; duration of hospitalization; the time to resolution of residual organ injury; and short-term (at 2 months of age) and long-term (at 1 year of age) survival. The primary endpoint will be the percentage of patients shedding virus (as detected by viral culture) from the oropharynx (i.e. throat) 5 days after beginning study drug. The secondary endpoints will include: duration (in days) of shedding of virus (as detected by viral culture) from the oropharynx, rectum, urine, and serum; change in baseline laboratory abnormalities [aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin, platelets, creatinine), reflecting either resolution or progression of enteroviral disease; pleconaril pharmacokinetics; safety; duration (in days) of total hospitalization; survival at 2 months of age; time (in days) to resolution of residual organ-related abnormalities following acute disease; and survival at 1 year of age.

ELIGIBILITY:
Inclusion Criteria:

-Signed informed consent statement by parent or legal guardian. -Age less than or equal to 15 days at time of onset of disease symptoms. Symptoms of systemic illness include but are not limited to fever, irritability, poor feeding, emesis, or diarrhea. Signs of systemic illness include, but are not limited to, jaundice, seizures, or lethargy. -Onset of disease symptoms less than or equal to 10 days (240 hours) prior to administration of first dose of study medication. -Birth weight greater than or equal to 1500 grams. -Gestational age of greater than or equal to 32 weeks. -Suspected or proven enteroviral disease. -One or more of the following three conditions: a. serum glutamic pyruvic transaminase (SGPT) greater than 3 times the upper limit of normal (ULN); b. platelet count less than 100,000 and prothrombin time greater than 1.5 times ULN and positive fibrin split products; c. cardiac shortening fraction less than 25% or cardiac ejection fraction less than 50% as measured by echocardiography.

Exclusion Criteria:

-Diagnosis of bacterial or non-enterovirus viral pathogen that can produce the constellation of presenting symptoms, known at the time of study enrollment. -Imminent demise (estimated life expectancy less than 24 hours). -Cyanotic congenital heart lesion. -Alimentary tract abnormalities which may interfere with the absorption of the study drug. These include mechanical obstruction of the gastrointestinal tract, necrotizing enterocolitis, and severe ileus (the definition of which is left to the clinical judgment of the participating investigator). -Infants known to be born to women who are human immunodeficiency virus (HIV) positive (but HIV testing is not required for study entry). These infants are at known risk of acquiring HIV, which would alter their immune response to other infections, including enteroviral infections. Additionally, they may be receiving antiretroviral and/or antiviral drugs during the time in which the study of pleconaril is being conducted. As such, they will be excluded if the mother's positive HIV status is known at the time of evaluation for study inclusion. If at any point following enrollment it is learned that an infant is HIV positive, however, he/she will be continued on the study protocol.

Ages: 0 Days to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2001-06-27 (Actual); Primary Completion 2010-09-22 (Actual); Study Completion 2012-09-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients shedding virus (as detected by viral culture) from the oropharynx (i.e. throat). | 5 days after beginning study drug.

SECONDARY OUTCOMES:
Change in baseline laboratory abnormalities [aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin, platelets, creatinine), reflecting either resolution or progression of enteroviral disease. | Day 1 (at study enrollment), 3, 5, 7, 10 and 14.
Duration (in days) of shedding of virus (as detected by viral culture) from the rectum, oropharynx (i.e. throat), urine and serum. | Day 1 (immediately prior to first dose of study drug), Days 2, 3, 4, 5, 7, 10 and 14.
Duration (in days) of total hospitalization. | At discharge from hospital.
Pleconaril pharmacokinetics. | Days 1, 3 and 7.
Safety. | After each clinical and safety evaluation during the treatment and follow-up period (through Day 180 +/- 14 days).
Survival at one year of age. | 1 year.
Survival at two months of age. | 2 months.
Time (in days) to resolution of residual organ-related abnormalities following acute disease. | Day(s) from onset of acute disease

CONTACTS AND LOCATIONS:
Locations (25):
- United States (24):
  - Children's of Alabama Child Health Research Unit (CHRU), Birmingham, Alabama
  - University of Arkansas - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Ronald Reagan University of California Los Angeles Medical Center, Los Angeles, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Stanford University - Stanford Hospital and Clinics - Pediatrics - Infectious Diseases, Stanford, California
  - Children's Hospital Colorado - Infectious Disease, Aurora, Colorado
  - University of Florida - Shands Children's Hospital, Gainesville, Florida
  - The University of Chicago - Comer Children's Hospital - Infectious Diseases, Chicago, Illinois
  - University of Louisville School of Medicine - Norton Children's Hospital - Infectious Diseases, Louisville, Kentucky
  - Tulane University - Tulane Medical Center - Pediatrics, New Orleans, Louisiana
  - University of Mississippi - Children's Infectious Diseases, Jackson, Mississippi
  - Washington University School of Medicine in St. Louis - Center for Clinical Studies, St Louis, Missouri
  - University of Nebraska Medical Center - Children's Hospital and Medical Center - Infectious Diseases, Omaha, Nebraska
  - Childrens Hospital at Saint Peters University Hospital - Allergy, Immunology and Infectious Diseases, New Brunswick, New Jersey
  - SUNY Upstate Medical University Hospital - Pediatrics, Syracuse, New York
  - Nationwide Children's Hospital - Infectious Diseases, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC - Allergy, Immunology and Infectious Diseases, Pittsburgh, Pennsylvania
  - Rhode Island Hospital - Pediatrics, Providence, Rhode Island
  - Vanderbilt University - Pediatric - Infectious Diseases, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center - Pediatrics, Dallas, Texas
  - Cook Children's Infectious Disease Services, Fort Worth, Texas
  - University of Texas Medical Branch - Pediatrics - Infectious Diseases and Immunology - Galveston, Galveston, Texas
  - University of Texas Health Science Center San Antonio - Pediatrics - Immunology & Infectious Disease, San Antonio, Texas
- University of Alberta Hospital - Pediatrics, Edmonton, Alberta, Canada